CLINICAL TRIAL: NCT04057508
Title: Effects of Non Invasive Vagus Nerve Stimulation on Heart Rate Variability in Healthy Subjects and on Muscle Sympathetic Nerve Activity
Brief Title: Non-invasive Modulation of Autonomic Cardiac Nervous System
Acronym: MSNA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université Catholique de Louvain (Other)
Collaborators: Erasme University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: TFE_201904_097
Record Dates: First submitted 2019-08-13; First posted 2019-08-15 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2019-07

CONDITIONS: Autonomic Nervous System; Heart Rate Variability; Muscle Sympathetic Nerve Activity
Keywords: Heart rate variability, MSNA, vagus nerve, sympathetic nervous system

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, double-blind, cross-over study
Who Masked: Participant, Investigator
Masking Description: Investigators are double-blinded for both experimental procedures and data analyzes.
  Volunteers are blinded to the site of stimulation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stimulation protocol (Active Comparator): Each subject will be blinded and underwent 3 phases of stimulation (actives (2) and sham (1) comparators) in a randomized order .
  Interventions: Other: Modulation of muscle sympathetic nerve activity
- Sham stimulation protocol (Sham Comparator): Each subject will be blinded and underwent 3 phases of stimulation (actives (2) and sham (1) comparators) in a randomized order.
  Interventions: Other: Modulation of muscle sympathetic nerve activity

INTERVENTIONS:
Other: Modulation of muscle sympathetic nerve activity — Assessment of muscle sympathetic nerve signal and exposition to external non invasive modulation.

SUMMARY:
To demonstrate the effect of non invasive vagus nerve (VNS) stimulation on heart rate variability and MSNA signal.

DETAILED DESCRIPTION:
First part: Assessment of the muscle sympathetic nerve activity (MSNA) at baseline using microneurography performed on the superficial peroneal nerve.

Second part: Acquisition of the MSNA signal during non-invasive VNS and apnea. Non-invasive VNS is performed using several frequencies of stimulation. Maximal and voluntaries apnea are performed at the end of the expiration.

Continuous recording of the following parameters:

* non-invasive arterial blood pressure
* R-R interval
* electrocardiogram
* MSNA activity
* respiratory curve signal
* respiratory rate, oxygen saturation

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* >18 years old

Exclusion Criteria:

* pregnancy and breastfeeding
* smoke
* alcool/energy drinks/coffee consumption, exertion 24h before the participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-06-19 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Heart rate variability modulation | 4 hours
  Modulation of heart rate variability assessed through analysis of MSNA signal

SECONDARY OUTCOMES:
Non-invasive vagus nerve stimulation | 4hours
  Modulation of parasympathetic tone based on two different frequencies stimulation
Profile of response for MSNA | 4 hours
  To describe positive and negative patterns of MSNA response

OTHER OUTCOMES:
Profile of response of MSNA during prolonged breath hold | 4hours
  Modulation of MSNA activity during repetitive prolonged breath hold

CONTACTS AND LOCATIONS:
Locations (1):
- Erasme University Hospital, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No